CLINICAL TRIAL: NCT06553274
Title: Effect of Nutritional Intervention Based on Predictive Model of Nutritional Factors on Survival of Adult Umbilical Cord Blood Transplantation Patients
Brief Title: Effect of Nutritional Intervention Based on Prediction Model on Adult Umbilical Cord Blood Transplantation Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nutrition-2024
Record Dates: First submitted 2024-08-05; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Nutrition Disorders
Keywords: umbilical cord blood transplantation; nutrition intervention
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Based on the nutritional factor prediction model, the individualized nutritional management of patients with umbilical cord blood transplantation (UCBT) was carried out to observe the impact on the survival efficacy of patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized nutrition intervention (Experimental): Full-time clinical nutrition pharmacists evaluate the nutritional status of enrolled patients and design individualized nutrition management programs
  Interventions: Procedure: Individualized nutrition intervention

INTERVENTIONS:
Procedure: Individualized nutrition intervention — After the patients were enrolled, they were given nutritional assessment by full-time clinical nutritionist and designed individualized nutritional management program, which included: Nutritional Assessment once a week for 4 weeks after Transplantation + 30 days, and nutritional assessment once a week for 4 weeks after Transplantation + 60 days, nutritional assessment every 2 weeks for 8 weeks; nutritional assessment every 4 weeks for 1 year after Transplantation + 120 days after transplantation; nutritional assessment during hospitalization in the ward and after discharge from the hospital, they were followed up in the nutrition counseling clinic or by telephone. The total energy intake was 25-35 kcal/kg/d and the protein intake was 1.2-1.5 g/kg/d. According to the"Five-step nutritional treatment principle", individual nutritional prescriptions were designed by clinical nutritionists.

SUMMARY:
Based on the nutritional factor prediction model, the individualized nutritional management of patients with umbilical cord blood transplantation (UCBT) was carried out to observe the impact on the survival efficacy of patients.

DETAILED DESCRIPTION:
The data of 80 UCBT patients were analyzed retrospectively, and the influence of nutritional parameters on the clinical outcome of UCBT patients was first confirmed, the skinfold thickness ≥20.5 mm and peripheral blood Alb < 33.6 g/L at 30 days after transplantation were the independent influencing factors of OS and DFS. In order to further verify the accuracy of the survival prediction model, the center intends to base on the model and aim at the nutritional parameters of patients 30 days after transplantation, a single-arm, single-center, phase II, prospective intervention trial was conducted to explore individualized nutrition management in UCBT patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, conscious, with language communication skills;
* UCBT patients to be performed;
* Major organs without serious dysfunction;
* The participants agreed to participate in the study and signed the informed consent form.

Exclusion Criteria:

* Age < 18 years old or > 65 years old or with cognitive impairment can not complete this survey;
* Failure or recurrence of transplantation;
* Combined with severe other organ system diseases (such as severe cardiac insufficiency, autoimmune disease, active infection, severe trauma) ;
* Patients who have difficulty collecting data to complete the nutritional intervention;
* Patients who asked to withdraw from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The body mass index | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  Body Mass Index (BMI) is defined as a person's weight in kilograms divided by the square of their height in meters (kg/m²).
The calf circumference | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  The calf circumference (cm)
The thickness of skinfold | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  thickness of skinfold (mm)
Grip strength | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  The grip strength (kg)
Prealbumin level | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  The level of prealbumin (mg/L)
Albumin Level | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  The level of Alb (g/L)

SECONDARY OUTCOMES:
Incidence of complications | before transplantation, Day30 , Day 60 , Day120 , Day180, 12 months after transplantation.
  Incidence of acute graft-versus-host disease (GVHD), incidence of chronic GVHD, incidence of oral mucositis and rate of infection.
Overall survival (OS) | 12 months after transplantation
  OS was calculated from the date of transplantation to death or last follow-up.
Disease-free survival (DFS) | 12 months after transplantation
  DFS was defined as the time from transplantation to relapse or death from any cause.
The cumulative incidence of relapse (CIR) | 12 months after transplantation
  Relapse and death were considered to be competing events when calculating CIR and NRM .
Non-Relapse Mortality (NRM) | 12 months after transplantation
  Relapse and death were considered to be competing events when calculating CIR and NRM .
Hospitalization Duration | 12 months after transplantation
  Hospitalization Duration
Hospitalization Costs | 12 months after transplantation
  expenses of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No